CLINICAL TRIAL: NCT06422611
Title: Comparison of Traditional and Digital Impression Methods for Pediatric Patients in Terms of Satisfaction
Brief Title: Comparing Dental Impression Methods for Children
Acronym: Digital
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Dilsah Cogulu, Professsor, Ege University
Other Study IDs: Ege U. Ethical Com. 23-4.1/5
Record Dates: First submitted 2024-02-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2023-04

CONDITIONS: Dental Impression, Pediatric Dentistry, Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Digital: Impression was taken with intraoral scanners
  Interventions: Device: Impression methods
- Conventional: Impression was taken with silicone impression material
  Interventions: Device: Impression methods

INTERVENTIONS:
Device: Impression methods — Both digital and conventional impressions were taken from same patients

SUMMARY:
The precision of dental restorations and the production of dental models has improved due to the acceleration of technical advancement and the introduction of computer-aided manufacturing.

The study's objective is to compare the conventional imprint approach with a digital one in order to compare patients' comfort levels, preferences, and treatment times among pediatric patients.

DETAILED DESCRIPTION:
In this study, 60 volunteers without any prior exposure to traditional or digital impressions took part. Using a C-type impression medium, conventional impressions of the maxillary and mandibular dental arches were taken. Digital impressions are taken using an intra-oral scanner at the same appointment. Following the impressions, a standardized questionnaire was used to assess the individuals' attitudes, preferences, and perceptions of the impression procedures. The Wong-Baker Pain Rating Scale was used to assess the perceived source of stress and Frankl Behavioural Scale was used for assessing behaviour. After taking the impression, the processing phases of the impression techniques (working time, etc.), and parental satisfaction were noted.

ELIGIBILITY:
Inclusion Criteria:

* not to have a history of digital or conventional impression taking
* not to have temporomandibular joint and periodontal discomfort
* not to be using psychiatric or neuropathic drugs

Exclusion Criteria:

* history of digital or conventional impression taking
* TMJ disorder
* Using any kind of drug that interferes pain perception

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients who needed routine diagnostic records were included in our study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Assessing patient preference and treatment comfort | March 2023-June 2023
  Parental satisfaction was measured with a structured questionnaire.The Wong-Baker Pain Rating Scale was used to assess the perceived source of stress and Frankl Behavioural Scale was used for assessing behaviour. A survey was designed to test 3 areas of patient satisfaction regarding the impression experience: comfort, time, and novelty. The survey consisted of 7 statements with a 100-mm visual analog scale (VAS) below each statement anchored with "agree" and "disagree." The survey also included questions to determine whether the patient had previous experience with impressions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No